CLINICAL TRIAL: NCT05442099
Title: The Effect of Iso-Principal Based Music Playlists on Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Frank Russo, Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB2020-068ISO2
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Anxiety State
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iso-principle music playlist (Experimental): Participants listen to the iso-principle music playlist for 30 minutes.
  Interventions: Behavioral: Iso-principle music playlist
- Generic calm music playlist (Sham Comparator): Participants listen to the generic music playlist for 30 minutes.
  Interventions: Behavioral: Generic calm music playlist

INTERVENTIONS:
Behavioral: Iso-principle music playlist — Participants listen to the iso-principle music playlist for 30 minutes.
  Arms: Iso-principle music playlist
Behavioral: Generic calm music playlist — Participants listen to the calm music playlist for 30 minutes.
  Arms: Generic calm music playlist

SUMMARY:
Chronic anxiety is a growing psychological challenge worldwide and at pre-clinical levels, can be disabling. Some research suggests music may reduce anxiety symptoms as effectively as anti-anxiety drugs without the adverse side effects. The iso principle suggests that the effectiveness of music interventions for mood management can be maximized by commencing a session with music that matches an individual's current emotional state and then gradually moving toward their desired emotional state. Our previous work demonstrated that a playlist generated by a music recommendation system that uses the iso-principal, along with music informatics, auditory beat stimulation, and reinforcement learning can reduce somatic and cognitive anxiety. However, it is unknown whether music playlists based on the iso-principal alone can reduce anxiety. In this study, the investigators wish to examine whether music playlists (~30 min long) based on the iso-principal (neutral to calm) will reduce anxiety after anxiety induction compared to a calm music playlist. The investigators hypothesize that the iso-principal playlist will have greater state anxiety reduction compared to the calm playlist.

DETAILED DESCRIPTION:
Chronic anxiety is a growing psychological challenge worldwide and at pre-clinical levels, can be disabling. Some research suggests music may reduce anxiety symptoms as effectively as anti-anxiety drugs without the adverse side effects. The iso principle suggests that the effectiveness of music interventions for mood management can be maximized by commencing a session with music that matches an individual's current emotional state and then gradually moving toward their desired emotional state. Our previous work demonstrated that a playlist generated by a music recommendation system that uses the iso-principal, along with music informatics, auditory beat stimulation, and reinforcement learning can reduce somatic and cognitive anxiety. However, it is unknown whether music playlists based on the iso-principal alone can reduce anxiety. In this study, the investigators wish to examine whether music playlists (~30 min long) based on the iso-principal (neutral to calm) will reduce anxiety after anxiety induction compared to a calm music playlist. The investigators hypothesize that the iso-principal playlist will have greater state anxiety reduction compared to the reverse-iso and calm playlists. Participants (n = 100) will be recruited and randomly assigned to one of three groups 1) Iso principal playlist, 2) Calm playlist. Prior to their treatment, all participants will undergo anxiety induction (recall an anxiety-provoking event, while listening to anxiety-inducing music). State anxiety (STICSA), positive and negative affect (PANAS), arousal, and valence (SAM) will be measured pre-post anxiety induction and after treatment. This work will be the first of its kind to examine whether a playlist based on the iso-principal is effective at reducing anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have no hearing impairments
* Participants who have no cardiac issues.
* Participants who have no history of seizures and epilepsy.

Exclusion Criteria:

* Participants who have hearing impairments
* Participants who have cardiac issues.
* Participants who have a history of seizures and epilepsy.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-08-15 (Estimated)

PRIMARY OUTCOMES:
Anxiety: State Trait Inventory for Cognitive and Somatic Anxiety (STICSA) | 30 minutes
  The STICSA has good reliability and validity as a measure of state and trait cognitive and somatic anxiety (Bados et al. 2010, Gros et al. 2007). The minimum score is 10 and the maximum is 40. Higher scores indicate higher anxiety (worse outcome). But in this study the post-intervention anxiety score is subtracted from the pre-intervention anxiety score, giving a measure of anxiety reduction. In the case of this anxiety reduction measure, higher anxiety reduction scores would indicate a better outcome.

SECONDARY OUTCOMES:
Mood: Positive and Negative Affect Scale (PANAS) | 30 minutes
  The PANAS has good reliability and validity and has been widely used in many studies to assess mood (Gray, 2007; Watson, Clark, & Tellegen, 1988). This scale generates two scores: 1) Positive affect (higher score indicates a better outcome), scores range from 10-50. 2) Negative affect (higher score indicates worse outcome), scores range from 10-50.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Russo, PhD, Principal Investigator — Toronto Metropolitan University; Adiel Mallik, PhD, Study Director — Toronto Metropolitan University

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data for STICSA state anxiety, PANAS, and SAM measures will be shared on the Open Science Framework.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available on the Open Science Framework (osf.io) when the pre-print of the study is uploaded to PsyArXiv. After that point the data will be available for a period of 5 years.
Access Criteria: All supporting information will be publicly accessible on the Open Science Framework (osf.io).

REFERENCES:
- [Background] Bados A, Gomez-Benito J, Balaguer G. The state-trait anxiety inventory, trait version: does it really measure anxiety? J Pers Assess. 2010 Nov;92(6):560-7. doi: 10.1080/00223891.2010.513295. PMID 20954057
- [Background] Davis WB, Thaut MH. The Influence of Preferred Relaxing Music on Measures of State Anxiety, Relaxation, and Physiological Responses. Journal of Music Therapy. 1989;26(4):168-87. doi: 10.1093/jmt/26.4.168.
- [Background] Gray EK, Watson, D. Assessing positive and negative affect via self-report. In: Coan JA, Allen, J.J.B., editor. Handbook of emotion elicitation and assessment. New York, NY: Oxford University Press; 2007.
- [Background] Gros DF, Antony MM, Simms LJ, McCabe RE. Psychometric properties of the State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA): comparison to the State-Trait Anxiety Inventory (STAI). Psychol Assess. 2007 Dec;19(4):369-81. doi: 10.1037/1040-3590.19.4.369. PMID 18085930
- [Background] Heiderscheit, A., & Madson, A. (2015). Use of the Iso Principle as a Central Method in Mood Management: A Music Psychotherapy Clinical Case Study. Music Therapy Perspectives, 33(1), 45-52. doi:10.1093/mtp/miu042 %J Music Therapy Perspectives
- [Background] Isik BK, Esen A, Buyukerkmen B, Kilinc A, Menziletoglu D. Effectiveness of binaural beats in reducing preoperative dental anxiety. Br J Oral Maxillofac Surg. 2017 Jul;55(6):571-574. doi: 10.1016/j.bjoms.2017.02.014. Epub 2017 Mar 18. PMID 28325532
- [Background] Mallik A, Russo FA. The effects of music & auditory beat stimulation on anxiety: A randomized clinical trial. PLoS One. 2022 Mar 9;17(3):e0259312. doi: 10.1371/journal.pone.0259312. eCollection 2022. PMID 35263341
- [Background] McConnell PA, Froeliger B, Garland EL, Ives JC, Sforzo GA. Auditory driving of the autonomic nervous system: Listening to theta-frequency binaural beats post-exercise increases parasympathetic activation and sympathetic withdrawal. Front Psychol. 2014 Nov 14;5:1248. doi: 10.3389/fpsyg.2014.01248. eCollection 2014. PMID 25452734
- [Background] Padmanabhan R, Hildreth AJ, Laws D. A prospective, randomised, controlled study examining binaural beat audio and pre-operative anxiety in patients undergoing general anaesthesia for day case surgery. Anaesthesia. 2005 Sep;60(9):874-7. doi: 10.1111/j.1365-2044.2005.04287.x. PMID 16115248
- [Background] Phillips SP, Yu J. Is anxiety/depression increasing among 5-25 year-olds? A cross-sectional prevalence study in Ontario, Canada, 1997-2017. J Affect Disord. 2021 Mar 1;282:141-146. doi: 10.1016/j.jad.2020.12.178. Epub 2020 Dec 30. PMID 33418360
- [Background] Starcke K, Mayr J, von Georgi R. Emotion Modulation through Music after Sadness Induction-The Iso Principle in a Controlled Experimental Study. Int J Environ Res Public Health. 2021 Nov 26;18(23):12486. doi: 10.3390/ijerph182312486. PMID 34886210
- [Background] Wahbeh H, Calabrese C, Zwickey H. Binaural beat technology in humans: a pilot study to assess psychologic and physiologic effects. J Altern Complement Med. 2007 Jan-Feb;13(1):25-32. doi: 10.1089/acm.2006.6196. PMID 17309374
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Yusim A, Grigaitis J. Efficacy of Binaural Beat Meditation Technology for Treating Anxiety Symptoms: A Pilot Study. J Nerv Ment Dis. 2020 Feb;208(2):155-160. doi: 10.1097/NMD.0000000000001070. PMID 31977827